CLINICAL TRIAL: NCT02645097
Title: Ideal Anatomic Location for Saphenous Nerve Blocks: A Prospective Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul J. Juliano, M.D. (Other)
Responsible Party: Sponsor-Investigator, Paul J. Juliano, M.D., Professor of Orthopaedic Surgery, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB - 39025
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Foot Injury; Ankle Injury
Keywords: Adult; nerve blocks in foot and ankle surgery; saphenous
MeSH Terms: conditions — Foot Injuries; Ankle Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal saphenous nerve block (Active Comparator): The anesthesiologist will administer a saphenous proximal nerve block if specified in the randomization envelope.
  Interventions: Procedure: Saphenous Nerve Block
- Distal saphenous nerve block (Active Comparator): The anesthesiologist will administer a saphenous distal nerve block if specified in the randomization envelope.
  Interventions: Procedure: Saphenous Nerve Block

INTERVENTIONS:
Procedure: Saphenous Nerve Block — A nerve block will be performed by the anesthesiologist. The location of the nerve block will be per randomization envelope (proximal vs. distal) and performed just prior to foot or ankle surgical procedures that require a saphenous nerve block

SUMMARY:
This research is being done to compare two different saphenous nerve block locations and will help to determine which site best maintains knee strength and pain control.

DETAILED DESCRIPTION:
This is a prospective, randomized, observer blinded clinical trial comparing motor strength in knee extension between two sets of patients, one receiving a proximal thigh block of the saphenous nerve and one receiving a distal thigh block of the saphenous nerve. The secondary objectives are to compare the pain relief and quality of life of participants in these two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Upcoming elective foot or ankle surgery

Exclusion Criteria:

* Preoperative weakness in knee extension
* Documented neuropathy
* Previous knee surgery
* Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
knee extensor strength measured in kilograms | change from baseline preoperatively to 30 minutes after nerve block placement
  Strength of the knee extensors in both treatment arms (distal vs. proximal block) will be tested preoperatively and again 30 minutes after the nerve block by using a hand-held dynamometer measured in kilograms

SECONDARY OUTCOMES:
pain level | change from baseline preoperatively to two weeks post-operatively
  Pain relief will be measured by review of the medical record for type and amount of pain medications used
quality of life assessment | change from baseline preoperatively to two weeks post-operatively
  PROMIS Global Health Survey will be completed by patients in both treatment arms pre-operatively and again two weeks post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Juliano, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No